CLINICAL TRIAL: NCT01513915
Title: A Parent-only Group Cognitive Behavioral Intervention for Children With Anxiety Disorders: a Control Waiting List Group Study
Brief Title: A Parent-only Group Cognitive Behavioral Intervention for Children With Anxiety Disorders: a Control Group Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Shahrivar, Assistant Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Parent CBT for Anxiety
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Anxiety Disorders
Keywords: parents; group cognitive behavioral intervention; anxiety disorder; children; FRIENDS program
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A parent only group CBT (Active Comparator): There was a Group cognitive behavioral intervention -based on parent training component of "FRIENDS" program- for parents of children with anxiety disorders who were allocated to intervention group.
  Interventions: Other: Group cognitive behavioral intervention
- Waiting list group (No Intervention): Parents of children with anxiety disorders who met the inclusion criteria and gave written informed consent and were allocated to wait list group.

INTERVENTIONS:
Other: Group cognitive behavioral intervention — A Group cognitive behavioral intervention _based on parent training component of FRIENDS program_ was performed.The program protocol was translated to Persian, using the back translation method.The intervention was delivered in 6 two-hour weekly sessions. Two intervention groups ran, each group included 10 parents.The therapy was provided by an attending board certified child and adolescent psychiatrist and co lead by a fellow of child and adolescent psychiatry who distributed psychometric procedures and completed treatment adherence ratings.
  Arms: A parent only group CBT

SUMMARY:
The fact that Cognitive Behavioral Therapy (CBT) is a well known efficacious intervention for children with anxiety disorders (AD) is undeniable. However, most children with AD have limited access to CBT. There is some controversial evidence on group CBT in AD involving families in treatment of their children and a published article on efficacy of a parent only group CBT for these children. Considering these data, the investigators hypothesized that teaching anxiety-fighting skills to parents of children with AD would diminish anxiety symptoms of both parents and children and improve family relational functioning.

DETAILED DESCRIPTION:
All children and their parents were interviewed using K-SADS-PL-Persian Version, a semi-structured diagnostic interview to confirm the diagnoses and assess possible comorbidities. All diagnostic assessments were conducted by a fellowship of child and adolescent psychiatry. Following assessment, once the participants reached twenty members, they were invited to complete child and parent self-report measures. The level of child functioning and family relationship functioning were also evaluated. Then they were randomly allocated to either parent training (N=20) or a 6 week wait-list (N=22) groups. During 2 weeks after treatment the assessments were repeated and satisfaction ratings were collected for the intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. having DSM-IV criteria for a primary diagnosis of generalized anxiety disorder (GAD), separation anxiety disorder (SAD), social phobia, or specific phobia.
2. age 6 to 12 years,
3. receiving one of selective serotonin reuptake inhibitor (SSRI) medicine at the stable dose for at least 8 weeks before baseline assessments and during the study,
4. at least one parent willing to participate and give written consent.

Exclusion Criteria:

1. diagnosed as bipolar disorder, autism spectrum disorders or mental disability by data obtained in personal history and clinical assessments,
2. there was a change in drug regime during the study period,
3. if parents missed more than 2 of 6 sessions of treatment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Revised Children's Manifest Anxiety (RCMA) | up to 30 minutes
  This self report questionnaire consists of 28 items assessing a child's chronic or trait anxiety and 9 items assessing social desirability or potential lying. The RCMA has achieved a high internal consistency and moderate test-retest reliability.

SECONDARY OUTCOMES:
Children's Depression Inventory (CDI) | 20 minutes
  This self report inventory has 27 items related to the cognitive, affective and behavioral signs of depression. The scale has high internal consistency and moderate test-retest reliability
Depression-Anxiety-Stress Scale (DASS) | 20 minutes
  This is a 42 item self-report instrument designed to measure the negative emotional states of depression, anxiety and stress. The DASS was shown to possess satisfactory psychometric properties.45-47 Parents completed this scale about their own negative emotional states
Children Global Assessment Scale (CGAS) | 15 minutes
  This Scale was developed to be a more child-specific measure of functioning. This measure is currently used in diagnosis, treatment, and evaluation of children's mental health problems to determine eligibility to receive mental health services and document treatment outcome status
Assessment of Consumer Satisfaction | 25 minutes
  Post treatment, parents in the intervention group completed a satisfaction questionnaire to rate how useful the program was in controlling their own anxiety, in managing their child anxious behavior, in improving family relations, the likelihood they would attend the treatment program again if needed, and if they would recommend the program to others on a 1 (not recommend) to 7 (highly recommend) likert scale
Strengths and Difficulties Questionnaire (SDQ) Home Version | [Time Frame: 30 minutes]
  This questionnaire is a parent report of psychopathology in children and adolescents. The scale consists of 25 items which generates five subscale scores (Emotional Symptoms, Conduct Problems, Inattention/Hyperactivity, Peer Problems and Prosocial Behavior) and a Total Difficulties Score. We used the SDQ Emotional Symptoms Scale (SDQ-Em) as a parent measure of child anxiety. SDQ has adequate internal consistency (α=0.37) and good test-retest reliability (r=0.62).42-44 The validity and reliability of SDQ has been confirmed in community samples of Iranian children and adolescents
Global Relational Assessment of Functioning (GRAF) | [Time Frame: 15 minutes]
  It provides a measure of the quality of functioning based on a review of three major areas: problem-solving, organization, and the emotional atmosphere. Available psychometric evidence suggests that clinician and even non clinician raters can achieve good to excellent reliability with only minimal training. The validity of the GRAF is supported by expected correlations with other measures of family and couple distress and functioning

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Shahrivar, MD, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Rouzbeh Hospital, Tehran, Tehran Province, Iran